CLINICAL TRIAL: NCT05670886
Title: Routine Bilateral Uterine Artery Ligation During the Cesarean Delivery of Multiple Gestation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassiony Dabian, lecturer of obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23BM73
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Postpartum Hemorrhage
Keywords: PPH - uterine artery ligation - carbetocin - multiple gesation
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- uterine artery ligation + carbetocin (Experimental): Group (A) , study group (N=55) : patients with multiple pregnancy undergoing cesarean section underwent bilateral uterine artery ligation and received carbetocin.
  Interventions: Procedure: uterine artery ligation
- carbetocin only (Active Comparator): Group (B ) , control group (N=55) : patients with twin pregnancy undergoing cesarean section received carbetocin only.
  Interventions: Procedure: uterine artery ligation

INTERVENTIONS:
Procedure: uterine artery ligation — The peritoneum over the vesico-uterine pouch already being incised horizontally, the peritoneum over the uterine isthmus and cervix was dissected downwards, and this dissection was then extended laterally Lower uterine incision was done followed by fetal extraction and placental delivery . bilateral uterine artery ligation were done 2cm below the uterine incision.
  Other Names: carbetocin

SUMMARY:
Multiple pregnancy is well defined to be associated with a greater risk of postpartum blood loss . Interventions to control PPH generally stepped from less to more invasive and including compression maneuvers , drugs , and further radical surgeries. Conservative management plans such as medications which cause the uterus to contract, external massage to the uterine body , and bimanual compression are overall used as 1st line interventions.

PPH was defined as a cumulative blood loss of 1,000 mL or more, or blood loss that occurred within 24 hours of childbirth and was accompanied by indications or symptoms of hypervolemia. The most frequent cause of PPH, which accounted for roughly 80% of cases, is uterine atony (3).

PPH is brought on by hyperexpansion, which impaired uterine myometrial contractility and caused uterine contraction fatigue , PPH were twice as high when pregnant with twins (4).The only effective surgical treatment for blood loss is a hysterectomy, but this is a risky procedure, especially for young women.(5)

Due to this, a number of fertility-preserving surgical procedures have been developed, including the B-Lynch technique, internal iliac artery ligation, and uterine artery ligation (UAL) One of the most widely used surgical methods for preserving fertility is UAL. It is simple to carry out and works well to control PPH. Additionally, it permits patients to have more children in the future and is generally safe. Additionally, it has a success rate of above 90%.

Concerns have been raised about its effect on women who want to become pregnant in the future regarding their ovarian reserve. The accepted practice of medicine worldwide is the prophylactic use of uterotonics. A synthetic oxytocin analogue with a lengthy half-life, carbetocin also stimulates uterine contractions .

One benefit of carbetocin over oxytocin is that it is more heat-stable, which is of greater importance to low resource settings . Studies compare the effectiveness of carbetocin and oxytocin in preventing PPH and find that carbetocin is equally effective or even more effective.

DETAILED DESCRIPTION:
This study is a randomized controlled study including a total number of 110 patients presenting to Kasr Al-ainy obstetrics and gynecology hospital for CS delivery. Ethical committee approved this study.

Patients are equally & randomly divided into two equal groups . Group (A) , study group (N=55) : patients with multiple pregnancy undergoing cesarean section undergoing bilateral uterine artery ligation and received carbetocin.

Group (B ) , control group (N=55) : patients with twin pregnancy undergoing cesarean section received carbetocin only.

Pregnant patients aging between 18 to 42 undergoing cesarean section for multiple pregnancy are included in this study , while Patients with Placenta previa or accrete , Ante-partum hemorrhage , patient refusing to participate , patients with medical disorders and patients with pre-operative HB less than 9 gm/dl were excluded from the study.

Informed consent was taken from involved patients after explanation of the procedures and their complications , and allocated patients were subjected to : (1) History taking regarding age , parity , previous CS , previous PPH , menstrual , medical and surgical history . (2) Examination : including general exam.(BMI , Blood Pressure ) , Abdominal examination ( Leopold's maneuvers , CS scars , fetal heart sounds , fundal level ) & local vaginal examination .

(3)Ultrasound was done to detect number of fetuses , gestational age , presentations , placental sites , amount of liquor & fetal weight. Patients were prepared for CS delivery after requesting pre-operative labs.

Anesthesia: spinal is mainly used except in cases were general anesthesia is indicated as fetal distress. Urinary catheterization and skin preparation was done. Skin incision using Pfannenstiel incision , opening abdomen in layers . The peritoneum over the vesico-uterine pouch already being incised horizontally, the peritoneum over the uterine isthmus and cervix was dissected downwards, and this dissection was then extended laterally Lower uterine incision was done followed by fetal extraction and placental delivery . Group (A): a single dose of 100 microgram carbetocin (Pabal® , ferring ) IV injection & bilateral uterine artery ligation were done 2cm below the uterine incision. Group (B): only a single dose of 100 microgram carbetocin (Pabal® , ferring ) IV injection administered after the delivery of the infant .

Closure of uterine incision & proper hemostasis were done . The abdomen was closed in layers . Patients were observed postpartum for vaginal bleeding , vitals , uterine tone , urine output & postoperative hemoglobin.

Operative time was calculated from the time of skin incision to tome of skin closure. Blood loss was calculated by Visual estimation by different operating room staff: the anesthetist, the obstetrician as well as the scrub nurse ( estimate the loss by careful observation of the operative field during surgery and report it at the end.) & by using weight of soaked towels (weight of soaked towel - weight of dry towel) and amount of blood in suction set. PPH was defined as blood loss of ≥1,000 ml following delivery (11).

Statistical Analyses were done using the Statistical Package for the Social Sciences (SPSS) , version 23. Quantitative Data were reported as mean± SD, while qualitative data were reported as number and percentage. The chi square test was used to compare categorical variables; P value <0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing cesarean section
* multiple pregnancy

Exclusion Criteria:

* Placenta previa.
* Ante-partum hemorrhage.
* patient refuse to participate

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant females with multiple gestations
Enrollment: 110 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-05 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
mean Blood loss after placental separation | 30 minutes
  by using weight of soaked towels (weight of soaked towel - weight of dry towel) and amount of blood in suction set

SECONDARY OUTCOMES:
Number of Participants with postpartum hemorrhage | 12 hours
  number pf participants with blood loss > 1000ml
The number of participant needed for blood transfusion | 24 hours
  Calculation of the number of participant needed for blood transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy outpatient infertility clinic, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 183: Postpartum Hemorrhage. Obstet Gynecol. 2017 Oct;130(4):e168-e186. doi: 10.1097/AOG.0000000000002351. PMID 28937571
- [Background] Santana DS, Cecatti JG, Surita FG, Silveira C, Costa ML, Souza JP, Mazhar SB, Jayaratne K, Qureshi Z, Sousa MH, Vogel JP; WHO Multicountry Survey on Maternal and Newborn Health Research Network. Twin Pregnancy and Severe Maternal Outcomes: The World Health Organization Multicountry Survey on Maternal and Newborn Health. Obstet Gynecol. 2016 Apr;127(4):631-641. doi: 10.1097/AOG.0000000000001338. PMID 26959199
- [Background] Gallos ID, Williams HM, Price MJ, Merriel A, Gee H, Lissauer D, Moorthy V, Tobias A, Deeks JJ, Widmer M, Tuncalp O, Gulmezoglu AM, Hofmeyr GJ, Coomarasamy A. Uterotonic agents for preventing postpartum haemorrhage: a network meta-analysis. Cochrane Database Syst Rev. 2018 Apr 25;4(4):CD011689. doi: 10.1002/14651858.CD011689.pub2. PMID 29693726
- [Background] Tulandi T, Sammour A, Valenti D, Child TJ, Seti L, Tan SL. Ovarian reserve after uterine artery embolization for leiomyomata. Fertil Steril. 2002 Jul;78(1):197-8. doi: 10.1016/s0015-0282(02)03164-3. No abstract available. PMID 12095516